CLINICAL TRIAL: NCT02928029
Title: A Phase 1b/2 Trial to Evaluate the Safety and Efficacy of Radium-223 Dichloride (BAY88-8223) in Combination With Bortezomib and Dexamethasone in Early Relapsed Multiple Myeloma
Brief Title: Study Testing Radium-223 Dichloride in Relapsed Multiple Myeloma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Due to the changes of standard of care and the slow recruitment of participants.
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18987; 2016-002438-58 (EudraCT Number)
Record Dates: First submitted 2016-10-06; First posted 2016-10-07 (Estimated); Results first posted 2020-02-26 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Multiple Myeloma
Keywords: Radium-223 dichloride; Bortezomib; Dexamethasone; Relapsed multiple myeloma; Combination therapy multiple myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — radium Ra 223 dichloride; Bortezomib; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase1, arm1: 33 kBq/kg Radium-223 dichloride+SOC (Experimental): Phase 1: Radium-223 dichloride; 33 kiloBecquerel (kBq)/kg body weight every 6 weeks for a total of 6 radium-223 dichloride doses plus SOC (standard of care) bortezomib/ dexamethasone.
  Interventions: Drug: Radium-223 dichloride (Xofigo, BAY88-8223); Drug: Bortezomib; Drug: Dexamethasone
- Phase1, arm2: 55 kBq/kg Radium-223 dichloride+SOC (Experimental): Phase 1: Radium-223 dichloride; 55 kBq/kg body weight every 6 weeks for a total of 6 radium-223 dichloride doses plus SOC bortezomib/ dexamethasone.
  Interventions: Drug: Radium-223 dichloride (Xofigo, BAY88-8223); Drug: Bortezomib; Drug: Dexamethasone
- Phase2, arm1: Placebo+SOC (Placebo Comparator): Phase 2: Matching placebo (isotonic saline) every 6 weeks for a total of 6 doses plus SOC bortezomib/dexamethasone.
  Interventions: Drug: Placebo; Drug: Bortezomib; Drug: Dexamethasone
- Phase2, arm2: Radium-223 dichloride+SOC (Experimental): Phase 2: Phase 1b-selected dose of radium-223 dichloride every 6 weeks for 6 doses plus SOC bortezomib/dexamethasone
  Interventions: Drug: Radium-223 dichloride (Xofigo, BAY88-8223); Drug: Bortezomib; Drug: Dexamethasone

INTERVENTIONS:
Drug: Radium-223 dichloride (Xofigo, BAY88-8223) — Sequential dose escalation in Intravenous (IV) injection
  Arms: Phase1, arm1: 33 kBq/kg Radium-223 dichloride+SOC; Phase1, arm2: 55 kBq/kg Radium-223 dichloride+SOC; Phase2, arm2: Radium-223 dichloride+SOC
Drug: Placebo — Matching placebo
  Arms: Phase2, arm1: Placebo+SOC
Drug: Bortezomib — Bortezomib is administered subcutaneous (SC) (per Investigator choice ) at 1.3 mg/m2/dose
Drug: Dexamethasone — Dexamethasone is administered orally at 40 mg

SUMMARY:
This study will be conducted in 2 parts. The phase 1b part will be an international, phase 1b, open-label, dose-escalation assessment of radium-223 dichloride administered with bortezomib and dexamethasone in subjects with relapsed multiple myeloma. The primary endpoint is to determine the optimal dose of radium-223 dichloride in combination with bortezomib/dexamethasone for the Phase 2 portion of the study.

The phase 2 part will be an international, phase 2, double-blind, randomized, placebo-controlled assessment of radium-223 dichloride versus placebo administered with bortezomib and dexamethasone, in subjects with relapsed multiple myeloma.

Up to 12 subjects in all dose cohorts combined will be treated in the phase 1b part of the study. Up to approximately 100 subjects will be enrolled in the phase 2 part of the study.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have documented monoclonal plasma cells in the bone marrow of ≥10%, as defined by their institutional standard at some point in their disease history or the presence of a biopsy proven plasmacytoma.
* Subjects must have received at least 1 and not more than 3 previous lines of treatment and have had a response to at least 1 prior Treatment in the past (i.e., achieved a minimal response [MR] or better) according to the IMWG uniform response criteria.
* Subject must be non-refractory to bortezomib (Refractory is defined: progression of disease while receiving bortezomib therapy or within 60 days of ending bortezomib therapy).
* Subjects must have documented evidence of progressive disease according to the IMWG uniform response criteria following the last multiple myeloma treatment.
* Subjects must have measurable disease defined as at least 1 of the following:

  * Serum M-protein defined by the following:

    * IgG multiple myeloma: Serum monoclonal paraprotein (M-protein) level ≥1.0 g/dL (measured by protein electrophoresis [PEP]);
    * IgA, IgD, IgE, IgM multiple myeloma: serum M-protein level ≥0.5 g/dL (measured by PEP).
  * Urine M-protein ≥200 mg/24 hours (any immunoglobulin heavy chain type measured by PEP).
  * Serum free light chain (FLC) ≥10 mg/dL with abnormal ratio in subjects with unmeasurable disease by serum or urine PEP.
* ≥1 bone lesion identifiable by radiograph, computed tomography (CT), positron emission tomography - computed tomography (PET-CT), or magnetic resonance imaging (MRI).
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0 to 2.
* Adequate hepatic function, with total bilirubin ≤1.5 x upper limit of normal (ULN) (except for Gilbert Syndrome: total bilirubin < 3.0 x ULN), and aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤3.0 x ULN.
* Absolute neutrophil count (ANC) ≥1.5 × 10e9/L, hemoglobin (Hb) ≥9.0 g/dL, and platelet count ≥75.0 × 10e9/L independent of transfusion of red blood cells (RBC) or platelet concentrates and independent of granulocyte colony-stimulating factor (G-CSF) or granulocyte-macrophage colony-stimulating factor (GM-CSF).
* International normalized ratio (INR) ≤ 1.5 and partial thromboplastin time (PTT) ≤ 1.5 x ULN. Prothrombin time (PT) may be used instead of INR if ≤ 1.5 x ULN.

Exclusion Criteria:

* Systemic glucocorticoid therapy (prednisone >10 mg/day orally or equivalent) within the last 4 weeks prior to first dose, unless tapered and on a stable dose (prednisone ≤10 mg/day orally or equivalent) for at least 1 week.
* Subjects with known POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes) or light-chain (AL) amyloidosis.
* Plasma cell leukemia (defined by plasma cell >20%, and/or an absolute plasma cell count of >2 x 10e9/L in peripheral blood).
* Subject has received anti-myeloma treatment within 2 weeks or 5 pharmacokinetic (PK) half-lives (t1/2) of the treatment, whichever is longer, before the date of start of treatment.
* Radiation therapy in the previous 4 weeks prior to first dose.
* Prior treatment with radium-223 dichloride or any experimental radiopharmaceutical.
* Congestive heart failure (New York Heart Association [NYHA] class III to IV), symptomatic cardiac ischemia, unstable angina or myocardial infarction in the previous 6 months prior to first dose, or with a known left ventricular ejection fraction (LVEF) <40%, cardiomyopathy, pericardial disease, clinically relevant cardiac arrhythmia (CTCAE version 4.03 Grade 2 or higher), clinically significant ECG abnormalities, or screening 12-lead ECG showing a baseline prolonged QT interval (baseline QT interval as corrected by Fridericia's formula > 470 msec).
* Neuropathy ≥ Grade 2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-02-10 (Actual); Primary Completion 2019-03-20 (Actual); Study Completion 2019-03-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (3):
  - Pacific Oncology/Hematology Associates, Encinitas, California
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- South Korea (2):
  - National Cancer Center, Goyang-si, Gyeonggido
  - Seoul National University Hospital, Seoul
- Spain (2):
  - Hospital Universitari Son Espases, Palma de Mallorca, Illes Baleares
  - Hospital Universitario Virgen del Rocío, Seville

REFERENCES:
- See also: Click here to find results for studies related to Bayer products — http://clinicaltrials.bayer.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 7 study centers, the first participant first visit was on 10/Feb/2017 and last participant last visit on 20/Mar/2019
Pre-assignment Details: 10 participants were screened in the study; 4 participants in Cohort 1 and 6 participants in Cohort 2. 3 of these participants failed screening procedures, all for the reason "inclusion criteria not met". No participants were started in the Phase 2 part of the study prior to study termination.
Groups:
- Radium-223 Dichloride 33 kBq/kg + Bortezomib and Dexamethasone: Participants received 33 kiloBecquerel (kBq)/kg body weight every 6 weeks for a total of 6 radium-223 dichloride doses in combination with BOR and DEX
- Radium-223 Dichloride 55 kBq/kg + Bortezomib and Dexamethasone: Participants received 55 kBq/kg body weight every 6 weeks for a total of 6 radium-223 dichloride doses in combination with BOR and DEX
Period: Overall Study
Arm/Group | Radium-223 Dichloride 33 kBq/kg + Bortezomib and Dexamethasone | Radium-223 Dichloride 55 kBq/kg + Bortezomib and Dexamethasone
Started | 3 | 4
Completed | 0 | 0
Not Completed | 3 | 4
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Radiological progression | 1 | 0
Not completed — Clinical progression | 1 | 2
Not completed — AE not related to clinical progression | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all randomized subjects who received at least one administration of study treatment
Groups:
- Total: Total of all reporting groups
Arm/Group | Radium-223 Dichloride 33 kBq/kg + Bortezomib and Dexamethasone | Radium-223 Dichloride 55 kBq/kg + Bortezomib and Dexamethasone | Total
Number analyzed (Participants) | 3 | 4 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.0 (5.0) | 68.3 (10.3) | 66.9 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 3 | 3 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 2 | 2
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Secondary Outcome: Phase 1: The Number of Subjects With Complete Response (CR) and Very Good Partial Response (VGPR)
Description: Determined by International Myeloma Working Group (IMWG) uniform response criteria.
  CR: Negative immunofixation of serum and urine, disappearance of any soft-tissue plasmacytomas, and <5% plasma cells in bone marrow; in patients for whom only measurable disease is by serum free light chain (FLC) level, normal FLC ratio of 0.26 to 1.65 in addition to CR criteria is required; 2 consecutive assessments are needed.
  VGPR: Serum and urine M-component detectable by immunofixation but not on electrophoresis or ≥90% reduction in serum M-component plus urine M-component <100 mg/24 hours (hrs); in patients for whom only measurable disease is by serum FLC level, >90% decrease in difference between involved and uninvolved FLC levels, in addition to VGPR criteria, is required; 2 consecutive assessments are needed
Time Frame: Up to approximately 2 years
Population: The safety analysis set including all participants who received at least one administration of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Radium-223 Dichloride 33 kBq/kg + Bortezomib and Dexamethasone | Radium-223 Dichloride 55 kBq/kg + Bortezomib and Dexamethasone
Number analyzed (Participants) | 3 | 4
Participants | NA — Participants were not evaluable per International Myeloma Working Group (IMWG) uniform response criteria | NA — Participants were not evaluable per International Myeloma Working Group (IMWG) uniform response criteria

2. Primary Outcome: Phase 1: MTD/RP2D Determined by the Incidence of DLTs
Description: Maximum tolerated dose (MTD) or recommended phase 2 dose (RP2D) determined by incidence of dose limiting toxicity (DLT) using Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 for the severity grade
Time Frame: From the start of study medication through 3 weeks after administration of the second dose of radium-223 dichloride, assessed up to 9 weeks
Population: The safety analysis set including all participants who received at least one administration of study treatment
Measure: Number; unit: KBq/kg
Arm/Group | Radium-223 Dichloride 33 kBq/kg + Bortezomib and Dexamethasone | Radium-223 Dichloride 55 kBq/kg + Bortezomib and Dexamethasone
Number analyzed (Participants) | 3 | 4
KBq/kg | NA — This study was stopped prior to the MTD being defined. Accordingly, there was no RP2D determined | NA — This study was stopped prior to the MTD being defined. Accordingly, there was no RP2D determined

3. Primary Outcome: Phase 1: The Number of Subjects With Treatment-emergent Adverse Events (TEAEs), Drug-related TEAEs, and Treatment-emergent Serious AE
Description: A treatment-emergent adverse event (TEAE) is defined as any event arising or worsening after start of study drug administration until the end of the treatment period
Time Frame: From the start of study drug (radium-223 dichloride) to 30 days after last dose of study treatment (radium-223 dichloride, BOR, or DEX, whichever is last), assessed up to approximately 2 years
Population: The safety analysis set including all participants who received at least one administration of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Radium-223 Dichloride 33 kBq/kg + Bortezomib and Dexamethasone | Radium-223 Dichloride 55 kBq/kg + Bortezomib and Dexamethasone
Number analyzed (Participants) | 3 | 4
Participants
  Any TEAE | 3 | 4
  Any drug-related TEAE | 3 | 4
  Any treatment-emergent serious AE | 2 | 1

ADVERSE EVENTS:
Time Frame: From the start of study drug (radium-223 dichloride) to 30 days after last dose of study treatment (radium-223 dichloride, BOR, or DEX, whichever is last), assessed up to approximately 2 years
Groups:
- Radium-223 33 kBq/kg + BOR/DEX: Subjects received 33 kiloBecquerel (kBq)/kg body weight every 6 weeks for a total of 6 radium-223dichloride doses in combination with BOR and DEX
- Radium-223 55 kBq/kg + BOR/DEX: Subjects received 55 kBq/kg body weight every 6 weeks for a total of 6 radium-223dichloride doses in combination with BOR and DEX
Arm/Group | Radium-223 33 kBq/kg + BOR/DEX | Radium-223 55 kBq/kg + BOR/DEX
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/4
Serious Adverse Events (participants affected / at risk) | 2/3 | 1/4
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radium-223 33 kBq/kg + BOR/DEX (N=3) | Radium-223 55 kBq/kg + BOR/DEX (N=4)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (4) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Spinal cord compression (Nervous system disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radium-223 33 kBq/kg + BOR/DEX (N=3) | Radium-223 55 kBq/kg + BOR/DEX (N=4)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (11)
Eye discharge (Eye disorders) | 0 (0) | 1 (1)
Eyelid oedema (Eye disorders) | 1 (1) | 0 (0)
Periorbital oedema (Eye disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 2 (2)
Visual acuity reduced (Eye disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (2) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 2 (4) | 2 (2)
Chest pain (General disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0)
Face oedema (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 2 (2)
Injection site reaction (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 2 (4) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (2) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Rhinovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Septic arthritis streptobacillus (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2)
Lymphocyte count decreased (Investigations) | 1 (3) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 2 (18)
Platelet count decreased (Investigations) | 0 (0) | 2 (16)
Weight decreased (Investigations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Hallucination (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 3 (3)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Nocturia (Renal and urinary disorders) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-09-28): https://cdn.clinicaltrials.gov/large-docs/29/NCT02928029/SAP_000.pdf
  • Study Protocol (2018-05-18): https://cdn.clinicaltrials.gov/large-docs/29/NCT02928029/Prot_001.pdf